CLINICAL TRIAL: NCT00621582
Title: Spiriva® 18µg Once Daily in Chinese COPD Patients of Different Disease Severities
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 205.373
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Results first posted 2010-06-15 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The objective of the present Post Marketing Surveillance Study (PMS) study is to evaluate safety and effectiveness of tiotropium bromide (Spiriva®) 18 µg once daily in 5,000 patients with COPD of varying severities over 8 weeks.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion Criteria:

Incl. Criteria Patients with clinical diagnosis of stable Chronic Obstructive Pulmonary Disease (COPD) according to definition of China COPD guideline.

Patients over 40 years old

Exclusion Criteria:

Patient with history of hypersensitivity to tiotropium bromide, atropine and/or its derivant, i.e. ipratropium, or any component of Spiriva® Patient with known narrow-angle glaucoma

* Patient with known symptomatic prostatic hyperplasia and/or bladder-neck obstruction
* Patient with known moderate to severe renal impairment (i.e.,creatinin clearance<=50ml/min)
* Pregnant or nursing women
* Patient with any significant disease other than COPD which would exclude him/her from participating in the study
* Patients with any conditions listed in [special precautions], [drug interactions], and [contraindication] of Spiriva® China package insert
* Patients with signed informed consent of any other study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 4918 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There is a gap between the enrollment number (4922) and the started patients (treatment number, 4812), as some of the enrolled patients did not accept the treatment.
  the number of started patients was 4918, among which 106 patients prematurely discontinued
Period: Overall Study
Arm/Group | Tiotropium Bromide
Started | 4918
Completed | 4812
Not Completed | 106
Not completed — Adverse Event | 7
Not completed — Protocol Violation | 57
Not completed — Lost to Follow-up | 24
Not completed — issues not identified by investigators | 18

BASELINE CHARACTERISTICS:
Arm/Group | Tiotropium Bromide
Number analyzed (Participants) | 4918
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (9.3)
Sex/Gender, Customized [Number; unit: participants]
  Female | 1603
  Male | 3313
  Missing information | 2

OUTCOME MEASURES:

1. Primary Outcome: Patient Global Assessment of Chronic Obstructive Pulmonary Disease (COPD) Symptom at Visit 1 and Visit 3 (Number of Patients Whose Assessment Were Excellent and Good)
Description: The score is evaluated according to a 8-point scale(poor: 1-2, fair: 3-4, good: 5-6, excellent: 7-8; 1 point meaning most COPD-associated symptoms and signs and 8 point meaning least).
  Represents number of participants who score ""good"" and ""excellent"" at visit 1 (0 weeks) and visit 3 (8 weeks)
Time Frame: 0 weeks (Visit 1) and 8 weeks (Visit 3)
Population: Sampling Method: Non-Probability Sample; conducted in primary care clinics.
Measure: Number; unit: Participants
Arm/Group | Tiotropium Bromide
Number analyzed (Participants) | 4918
Participants
  Number of patients at visit 1 | 831
  Number of patients at visit 3 | 4213
Statistical Analysis 1: Comparison: Tiotropium Bromide; comparing results of post-treatment global assessment by patient with that of pre-treatment; Test type: Superiority or Other; p = 0.01, Chi-squared

2. Secondary Outcome: Physician Global Assessment of Spiriva Effectiveness at Visit 2 and Visit 3 (Number of Patients Whose Assessment Were Excellent and Good)
Description: The score is evaluated according to a 8-point scale(poor: 1-2, fair: 3-4, good: 5-6, excellent: 7-8;
  Represents number of participants who score ""good"" and ""excellent"" at visit 2 (2 weeks) and visit 3 (8 weeks)
Time Frame: 2 weeks (Visit 2 and 8 weeks (Visit 3)
Measure: Number; unit: Participants
Arm/Group | Tiotropium Bromide
Number analyzed (Participants) | 4918
Participants
  Number of patients at visit 2 | 4005
  Number of patients at visit 3 | 4694

3. Primary Outcome: Patient Tolerability Assessment at Visit 3
Description: Patient tolerability assessment classified as "Unsatisfied", "Satisfied", "Good" and "Very Good"
Time Frame: 8 weeks (Visit 3)
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Tiotropium Bromide
Number analyzed (Participants) | 4880
Participants
  Unsatisfied | 5
  Satisfied | 196
  Good | 1570
  Very Good | 3109

4. Secondary Outcome: Physician Tolerability Assessment at Visit 3
Description: The score is evaluated according to a 8-point scale(poor: 1-2, fair: 3-4, good: 5-6, excellent: 7-8)
Time Frame: 8 weeks (Visit 3)
Population: Full Analysis Set (FAS)
Measure: Number; unit: Participants
Arm/Group | Tiotropium Bromide
Number analyzed (Participants) | 4880
Participants
  Poor | 2
  Fair | 90
  Good | 1112
  Excellent | 3676

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Tiotropium Bromide
Serious Adverse Events (participants affected / at risk) | 4/4918
Other Adverse Events (participants affected / at risk) | 0/4918
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium Bromide (N=4918)
Exacerbation of chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Acute pancreatitis (Gastrointestinal disorders) | 1
Acute heart failure (Cardiac disorders) | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Shock (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.